CLINICAL TRIAL: NCT05602233
Title: The Effect of Balance Training Following STARS on Postural Control and Function in Athletes With Chronic Ankle Instability
Brief Title: The Effect of Balance Training Following STARS on Postural Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ankle-BAU&HBU-20221012
Record Dates: First submitted 2022-10-26; First posted 2022-11-02 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Kinesiophobia; Ankle Sprains; Sensory Deficit; Ankle Instability; Functional Performance
MeSH Terms: conditions — Kinesiophobia; Ankle Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants between the ages of 18-25, diagnosed with chronic ankle sprain who met the inclusion criteria will be included in the study. Sample size of the study is calculated as 21. All evaluations of the participants, including postural control, weight bearing dorsiflexion angle measurement, function and kinesiophobia will be made by the same physiotherapist. The physiotherapist who made the evaluations will not know which treatment method will be applied to the participants.
Who Masked: Outcomes Assessor
Masking Description: The physiotherapist who made the evaluations will be blind to the groups. He will not know which treatment method will be applied to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Balance training: (Experimental): It is planned to apply hop to stabilization exercises developed by Mckeon et al. The training will be given for 6 weeks, 3 times a week for 20 minutes. This phased balance training program is based on the participant's ability to maintain a single limb posture while performing balance activities. The program includes: 1) hop to stabilization, 2) hop to stabilization and reach, 3) hop to stabilization box drill, 4) progressive single-limb stance balance activities with eyes open, and 5) progressive single-limb stance activities with eyes closed. Participants will be followed up with a physiotherapist and will be able to proceed to the next stage of the test after completing the previous level without errors.
  Interventions: Other: Exercise
- STARS (Experimental): A combination of STARS developed by Mckeon et al. is planned for the STARS group. The training will be given for 6 weeks, 3 times a week for 5 minutes. STARS includes; joint mobilization, plantar massage and triceps surae stretching.
  Interventions: Other: STARS (Sensory-Targeted Ankle Rehabilitation Strategies)
- Combined Training (Experimental): Each participant in the combined training program will receive 4 weeks of balance training after 2 weeks of STARS treatment. STARS and hop to stabilization treatment protocol will be applied in the same way.
  Interventions: Other: Exercise; Other: STARS (Sensory-Targeted Ankle Rehabilitation Strategies)

INTERVENTIONS:
Other: Exercise — The training will be given for 6 weeks, 3 times a week for 20 minutes. This phased balance training program is based on the participant's ability to maintain a single limb posture while performing balance activities. The program includes: 1) hop to stabilization, 2) hop to stabilization and reach, 3) hop to stabilization box drill, 4) progressive single-limb stance balance activities with eyes open, and 5) progressive single-limb stance activities with eyes closed. Participants will be followed up with a physiotherapist and will be able to proceed to the next stage of the test after completing the previous level without errors.
  Arms: Balance training:; Combined Training
Other: STARS (Sensory-Targeted Ankle Rehabilitation Strategies) — STARS includes; joint mobilization, plantar massage and triceps surae stretching. The training will be given for 6 weeks, 3 times a week for 5 minutes.
  Arms: Combined Training; STARS

SUMMARY:
Chronic ankle instability (CAI) is defined as the symptoms continuing 12 months after the first sprain and the functional and/or mechanical instability reported by the individual. The number of researches that include a combined treatment approach that will affect both sensory and motor components in rehabilitation strategies applied for CAI is limited.

The aim of this study is to isolated sensory, isolated motor and combined targeted approaches for the treatment of chronic ankle instability (CAI); to compare the effects on postural control, range of motion, function and kinesiophobia and to contribute to an effective approach related to the applicability of Sensory-Targeted Ankle Rehabilitation Strategies in the treatment of CAI.

DETAILED DESCRIPTION:
Lateral ankle sprains are among the most common injuries in athletes and physically active individuals, accounting for 80% of ankle injuries. After the ankle is sprained for the first time, it becomes more prone to re-injury. Chronic ankle instability (CAI) is defined as the symptoms continuing 12 months after the first sprain and the functional and/or mechanical instability reported by the individual. Long-term ongoing CAI symptoms; It includes pain, swelling, give away that reduces the person's quality of life.

Symptoms of CAI include both motor and sensory aspects of the sensorimotor system. Despite sensory and motor deficits in sensorimotor control, researches on CAI rehabilitation have focused on either motor or sensory components. The number of researches that include a combined treatment approach that will affect both sensory and motor components in rehabilitation strategies applied for CAI is limited.

Sensory-Targeted Ankle Rehabilitation Strategies (STARS) and balance training have proven to be effective in relieving CAI-associated deficits. Although the effects of isolated STARS were positive, in a recent study, there was no statistically significant difference between the groups when the balance training given with STARS was compared with the balance training alone. However, the reason for the lack of difference between the groups may be the simultaneous application of both treatment protocols. In addition, the effects of the isolated use of the STARS combination in the treatment of CAI are still unclear and to our knowledge, there are no studies in this area.

The aim of this study is to isolated sensory, isolated motor and combined targeted approaches for the treatment of chronic ankle instability (CAI); to compare the effects on postural control, range of motion, function and kinesiophobia and to contribute to an effective approach related to the applicability of STARS in the treatment of CAI.

ELIGIBILITY:
Inclusion Criteria:

* History of first ankle sprain more than 1 year ago

  * Having at least 2 "give away" episodes in the last 6 months
  * Identification of Functional Ankle Instability's score above 11
  * 18-25 age range
  * Foot and Ankle Ability Measure (FAAM), the score of which is less than %90
  * Foot and Ankle Ability Measure Sports scale (FAAM-S), the score of which is less than %80

Exclusion Criteria:

* History of lower extremity surgery
* History of disease that may affect sensorimotor function in the lower extremity
* Musculoskeletal disorders that may affect balance

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Postural control evaluation change | Change from Baseline postural control at 6 weeks
  Star excursion balance test (SEBT): The star excursion balance test is frequently used to evaluate the dynamic balance and postural control of the lower extremities. SEBT, is a test that measures the maximum reach of the individual by maintaining balance and performing a single-leg squat in lines drawn at 45 degrees intervals in eight different directions. The participant stands in the middle of the star shape with bare feet. For the starting position, the ankle should be stationary, the hands on the hips, and the participant should maintain the starting position throughout the test. The participant is asked to reach anteriorly, posteromedially and posterolaterally with the unstable ankle, make a light touch to the line, and rotate the outstretched leg back to the center while maintaining a one-leg stance with the other leg.The participant will be allowed to make 4 trials in each direction

SECONDARY OUTCOMES:
Ankle dorsiflexion measurement change | Change from baseline ankle dorsiflexion measurement at 6 weeks
  Weight-bearing lunge test (WBLT) is frequently used in individuals with ankle instability in order to determine dorsiflexion normal joint movement. During WBLT the participant puts his hands on the wall and takes one leg forward and the other leg helps balance behind. The maximum distance that the knee touches the wall is recorded without allowing the heel of the front foot to lose contact with the ground.
Function change | Change from baseline ankle function measurement at 6 weeks
  The Foot and Ankle Ability Measure is used to assess self-reported overall function levels in patients with leg, ankle, and foot musculoskeletal injuries and disorders. It consists of 2 subscales (Activities of Daily Living [ADL] and Sports [S]), both scored between 0% and 100%. The FAAM-ADL is a 21-item scale to assess function during activities of daily living. FAAM-Sport is an 8-item scale focusing on sports-related activities. Items in both tools are scored on a 5-point Likert scale ranging from 0 (no difficulty at all) to 4 (I can't do it). Scores are converted to percentages, and a higher percentage indicates a better level of function.
Kinesiophobia change | Change from baseline kinesiophobia measurement at 6 weeks
  The Tampa kinesiophobia scale is often used in musculoskeletal injuries. TKS has a checklist of 17 questions. A 4-point Likert scoring (1= I strongly disagree, 4= I totally agree) is used in the scale. After reversing items 4, 8, 12 and 16, a total score is calculated. The person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PhD, PT, Study Chair — Bahçeşehir University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Serkan Uzlaşır, PhD, PT, Study Director — Nevsehir Haci Bektas Unıversity, Faculty of Sports Sciences, Department of Coaching Education; Aynur Merve Zümre, PT, Principal Investigator — Bahçeşehir University, Graduate Education Institute, Physical Therapy and Rehabilitation Program
Locations (1):
- Bahcesehir University, Beşiktaş, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No